CLINICAL TRIAL: NCT07319676
Title: Antigen Targeted T Cell Therapy for Relapsed/Refractory B Cell Lymphomas
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022/00272
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-09

CONDITIONS: B-cell Lymphoma Refractory
Keywords: Antigen targeted; T cell therapy; Relapsed/Refractory B cell lymphomas
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: This study will start with the phase 1 lead in to determine the R2PF followed by a phase 2 trial to evaluate the safety and efficacy of Epo-R-CD19 CAR T with or without CD22 CAR T-cells infused into patients with BCL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR T-cells (Experimental): The CAR T-cells used in this clinical trial are autologous T cells that have been cultured ex vivo and transduced with a retroviral vector delivering a gene encoding a CAR, as described in the accompanying Chemistry, Manufacturing and Controls (CMC) document.
  Each infusion bag will have affixed to it a label containing the following: product identifier, product name and volume. In addition, the label will also have at least 2 unique identifiers such as name of patient, patient's alphanumeric identifier and birth date, according to applicable regulations. Prior to infusion, 2 individuals will verify all information and confirm the identity to ensure that the information is correctly matched to the patient and that the patient receives only their autologous product. This is done according to local institutional guidelines.
  Interventions: Other: CART infusion

INTERVENTIONS:
Other: CART infusion — CART cells originate with the isolation of the patient's T cells via apheresis. These cells are then activated and modified to express a transgene that encodes a tumor-specific CAR. These cells are then expanded to achieve a clinically significant cell dose which will then be infused back into the patient. After CART infusion, these CART cells will come into contact with the tumor-specific antigen on the surface of the tumor cells, activating the CART cells which will expand and kill the tumor cells.

SUMMARY:
This is a single center, open label, phase 1 lead in to determine Recommended Phase 2 Dose (RP2D), followed by a phase 2 trial to evaluate the safety and efficacy of Epo-R-CD19 CAR T with or without CD22 CAR T-cells infused into patients with B cell lymphoma.

The study will have the following parts:

* Screening
* Pre-infusion (cell product preparation and bridging) and infusion (lymphodepletion)
* Primary efficacy endpoints
* Long term follow up

Patients who have high risk B cell lymphoma or relapsed/refractory B cell lymphoma who fufil the trial inclusion and exclusion criteria will undergo leukapheresis following trial enrollment.

CAR T-cell products will then be manufactured according to the antigen expression on the patient's biopsied tumor cells. These cells will then undergo stringent testing before the patient undergoes lymphodepletion followed by CART infusion. These patients will be admitted for the infusion and closely monitored for any CRS or ICANS.

This study will have a Phase 1 safety run in for the first 3-6 patients who receive the Epo-R-CD19 CAR T (with or without epoetin (erythropoietin)) to determine the tolerability and safety of this product. For the first 3-6 patients, if there are any DLT seen by Day 28, a data safety monitoring committee will be convened to assess the trial. Staggered dosing will be implemented for the first 2 participants in every dose level (DL1, DL2 and DL-1).

For Phase 2, the RP2D will depend on DLT. If there is no DLT at DL+1 and DL+2, then the investigators will proceed with DL+2 as the RP2D dose. On the other hand, if there is DLT despite DL-1, then the study will be redesigned. Phase 2 will continue until a total of 20 patients received their CAR T-cell infusions.

CAR-T monitoring will be performed at Day 0, 7, 14, 21, 28, month 2, 3, 4, 5, 6, 12 and yearly thereafter. The total duration of the study is 15 years from CAR T infusion.

DETAILED DESCRIPTION:
2.1 Hypothesis

1. The infusion of CD19 with or without CD 22 targeted CAR T-cells in patients with high risk or R/R BCL will improve the overall response rates and survival outcomes. The choice of antigen target is determined by detailed flow cytometric profiling of biopsied lymphoma cells if possible.
2. The co-expression of Epo-R in our CD19 CAR T-cells will allow endogenous or exogenous Epo levels to support survival and expansion of infused T cells, thus overcoming the issue of suboptimal T-cell expansion and persistence due to prior chemotherapies in patients with high risk or R/R DLBCL.

2.2 Objectives for Phase 1:

Primary objective of Phase 1 lead in is to determine safety, as defined by incidence of dose limiting toxicities (DLT) associated to the Epo-R-CD19 CAR and CD22 pooled products, as well as determination of the RP2D of the Epo-R-CD19

The secondary objective is to assess efficacy of the Epo-R-CD19 CAR as defined by:

i) Percentage of patients who achieve peak CAR T level within Month 1 > 30 CD 19 CAR-T cells/uL ii) Proportion of patients who achieved no evidence of disease as determined PET-CT using the Lugano criteria at 1 month and the best overall response by 6 months as assessed by PET-CT (Lugano criteria).

2.3 Objectives For Phase 2:

The primary objective of Phase 2 is efficacy. The primary endpoints are:

a. To determine the efficacy of a single Epo-R-CD19 CAR T-cell or a pool of CAR T-cells targeting CD19 and CD22 antigens based on detailed flow cytometric profiling of high risk or R/R BCL patients. The efficacy is determined by the proportion of patients who achieved no evidence of disease as determined PET-CT using the Lugano criteria at 1 month and the best overall response by 6 months as assessed by PET-CT (Lugano criteria).

Our secondary endpoints are:

1. To determine the safety of the Epo-R-CD19 and CD22. The investigators will collect data on CAR T related toxicities: This includes incidence of dose limiting toxicities (Section 5), treatment related adverse events (Section Table 4.9) and adverse events of special interest (Section 2.5).
2. To determine the peripheral blood levels of CAR CD19 and CD22 at D0, D5, D7, D14, D21 and 1 month, 3 months, 6 months, 1 year and 2 years. The investigators will compare our Epo-R-CD19 CAR T-cell levels against CD22 and published commercial CAR T expansion.
3. To study the 1-year Event free survival defined by any event involving disease recurrence or persistence disease at 6 months, death from any cause. Planned HSCT, after CAR T infusion, is not an event
4. To study the 1-year Overall Survival
5. Cumulative risk of relapse (CIR), defined as proportion of patients surviving 1-year after CAR T-cell infusion.

ELIGIBILITY:
Inclusion Criteria

* Age 10 to 80 years at screening
* PET-CT measurable disease by Lugano classification (Deauville score of ≥4) and
* Tissue biopsy of any tumour site and flow cytometry study of CD19 and CD22 expression.
* Relapsed B-cell lymphoma after one line of systemic therapy or autologous bone marrow transplant. This includes DLBCL, PMBCL, HGBCL, DLBCL arising from indolent lymphoma, Burkitt's lymphoma/leukemia, Mantle cell lymphoma.
* High risk B-cell lymphoma (BCL). High risk BCL is defined by any of the criteria below:

  * High-risk genetics - double/triple hit or p53mut or deletion.
  * IPI score ≥ 3
  * Richter's transformation from chronic lymphocytic leukaemia.
  * Disease refractory to treatment - PET-CT positive disease after 2 courses of rituximab-containing chemoimmunotherapy.
* PBMC product available
* Karnofsky or Lansky score >70. Or ECOG 0-2
* Patient expected survival is more than 3 months to allow for manufacture and release of CAR T-cells.

Exclusion Criteria

* Patients who test positive on urine or blood pregnancy testing and are pregnant or are lactating.
* Participant of reproducible age who refuse the use of the following birth control methods if engaging in sexual activity that could lead to pregnancy. The methods include condoms, diaphragm, intrauterine device, hormonal based contraception.
* Concomitant genetic syndromes associated with BM failure states, such as Fanconi anaemia, Kostmann syndrome, Schwachman syndrome, or any other BM failure syndrome with the exception of Down syndrome.
* Active hepatitis B or hepatitis C within 3 months of screening.
* Active HIV infection within 3 months of screening.
* Grade 2 to 4 graft-vs-host disease (GVHD).
* Received an investigational medicinal product within 1 month of screening.
* If the total sum of CD19 and CD22 antigens expressed is less than 95.0%, patients will not be eligible. If subsequent immunophenotying of the patient's sample confirms that total sum of CD19 and CD22 antigens ≥ 95%, the patient may be rescreened.
* Central nervous system: Uncontrolled seizures or status epilepticus; decreased conscious state (any cause)
* Foreign patients who cannot commit to agreeable to stay in Singapore for at least 3 months post CAR T infusion and are committed to the long term monitoring post CAR T at home and in Singapore.
* Prior treatment with any CAR T cell therapy (approved or investigational)

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2040-10-31 (Estimated)

PRIMARY OUTCOMES:
Best objective response post CAR-T infusion | 6 months
  Best objective response will be assessed using standardised lymphoma response criteria at regular intervals up to 6 months post CAR-T infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Poon, Principal Investigator — NUHS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee DW, Gardner R, Porter DL, Louis CU, Ahmed N, Jensen M, Grupp SA, Mackall CL. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014 Jul 10;124(2):188-95. doi: 10.1182/blood-2014-05-552729. Epub 2014 May 29. PMID 24876563
- [Result] Neelapu SS, Tummala S, Kebriaei P, Wierda W, Gutierrez C, Locke FL, Komanduri KV, Lin Y, Jain N, Daver N, Westin J, Gulbis AM, Loghin ME, de Groot JF, Adkins S, Davis SE, Rezvani K, Hwu P, Shpall EJ. Chimeric antigen receptor T-cell therapy - assessment and management of toxicities. Nat Rev Clin Oncol. 2018 Jan;15(1):47-62. doi: 10.1038/nrclinonc.2017.148. Epub 2017 Sep 19. PMID 28925994
- [Result] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Result] Garcia Borrega J, Godel P, Ruger MA, Onur OA, Shimabukuro-Vornhagen A, Kochanek M, Boll B. In the Eye of the Storm: Immune-mediated Toxicities Associated With CAR-T Cell Therapy. Hemasphere. 2019 Mar 29;3(2):e191. doi: 10.1097/HS9.0000000000000191. eCollection 2019 Apr. PMID 31723828
- [Result] Gisselbrecht C, Glass B, Mounier N, Singh Gill D, Linch DC, Trneny M, Bosly A, Ketterer N, Shpilberg O, Hagberg H, Ma D, Briere J, Moskowitz CH, Schmitz N. Salvage regimens with autologous transplantation for relapsed large B-cell lymphoma in the rituximab era. J Clin Oncol. 2010 Sep 20;28(27):4184-90. doi: 10.1200/JCO.2010.28.1618. Epub 2010 Jul 26. PMID 20660832
- [Result] Crump M, Neelapu SS, Farooq U, et al. Outcomes in refractory diffuse large B-cell lymphoma: results from the international SCHOLAR-1 study. Blood. 2017;130(16):1800-1808. Blood. 2018 Feb 1;131(5):587-588. doi: 10.1182/blood-2017-11-817775. No abstract available. PMID 29437609
- [Result] Schuster SJ, Bishop MR, Tam CS, Waller EK, Borchmann P, McGuirk JP, Jager U, Jaglowski S, Andreadis C, Westin JR, Fleury I, Bachanova V, Foley SR, Ho PJ, Mielke S, Magenau JM, Holte H, Pantano S, Pacaud LB, Awasthi R, Chu J, Anak O, Salles G, Maziarz RT; JULIET Investigators. Tisagenlecleucel in Adult Relapsed or Refractory Diffuse Large B-Cell Lymphoma. N Engl J Med. 2019 Jan 3;380(1):45-56. doi: 10.1056/NEJMoa1804980. Epub 2018 Dec 1. PMID 30501490
- [Result] Locke FL, Ghobadi A, Jacobson CA, Miklos DB, Lekakis LJ, Oluwole OO, Lin Y, Braunschweig I, Hill BT, Timmerman JM, Deol A, Reagan PM, Stiff P, Flinn IW, Farooq U, Goy A, McSweeney PA, Munoz J, Siddiqi T, Chavez JC, Herrera AF, Bartlett NL, Wiezorek JS, Navale L, Xue A, Jiang Y, Bot A, Rossi JM, Kim JJ, Go WY, Neelapu SS. Long-term safety and activity of axicabtagene ciloleucel in refractory large B-cell lymphoma (ZUMA-1): a single-arm, multicentre, phase 1-2 trial. Lancet Oncol. 2019 Jan;20(1):31-42. doi: 10.1016/S1470-2045(18)30864-7. Epub 2018 Dec 2. PMID 30518502
- [Result] Viardot A, Goebeler ME, Hess G, Neumann S, Pfreundschuh M, Adrian N, Zettl F, Libicher M, Sayehli C, Stieglmaier J, Zhang A, Nagorsen D, Bargou RC. Phase 2 study of the bispecific T-cell engager (BiTE) antibody blinatumomab in relapsed/refractory diffuse large B-cell lymphoma. Blood. 2016 Mar 17;127(11):1410-6. doi: 10.1182/blood-2015-06-651380. Epub 2016 Jan 11. PMID 26755709
- [Result] Stirrups R. CAR T-cell therapy for relapsed or refractory mantle-cell lymphoma. Lancet Oncol. 2020 May;21(5):e239. doi: 10.1016/S1470-2045(20)30231-X. Epub 2020 Apr 9. No abstract available. PMID 32278358
- [Result] Fry TJ, Shah NN, Orentas RJ, Stetler-Stevenson M, Yuan CM, Ramakrishna S, Wolters P, Martin S, Delbrook C, Yates B, Shalabi H, Fountaine TJ, Shern JF, Majzner RG, Stroncek DF, Sabatino M, Feng Y, Dimitrov DS, Zhang L, Nguyen S, Qin H, Dropulic B, Lee DW, Mackall CL. CD22-targeted CAR T cells induce remission in B-ALL that is naive or resistant to CD19-targeted CAR immunotherapy. Nat Med. 2018 Jan;24(1):20-28. doi: 10.1038/nm.4441. Epub 2017 Nov 20. PMID 29155426
- [Result] Pasquini MC, Hu ZH, Curran K, Laetsch T, Locke F, Rouce R, Pulsipher MA, Phillips CL, Keating A, Frigault MJ, Salzberg D, Jaglowski S, Sasine JP, Rosenthal J, Ghosh M, Landsburg D, Margossian S, Martin PL, Kamdar MK, Hematti P, Nikiforow S, Turtle C, Perales MA, Steinert P, Horowitz MM, Moskop A, Pacaud L, Yi L, Chawla R, Bleickardt E, Grupp S. Real-world evidence of tisagenlecleucel for pediatric acute lymphoblastic leukemia and non-Hodgkin lymphoma. Blood Adv. 2020 Nov 10;4(21):5414-5424. doi: 10.1182/bloodadvances.2020003092. PMID 33147337
- [Result] Chow VA, Gopal AK, Maloney DG, Turtle CJ, Smith SD, Ujjani CS, Shadman M, Cassaday RD, Till BG, Tseng YD, Warren EH, Shustov AR, Menon MP, Bhark S, Acharya UH, Mullane E, Hannan LM, Voutsinas JM, Gooley TA, Lynch RC. Outcomes of patients with large B-cell lymphomas and progressive disease following CD19-specific CAR T-cell therapy. Am J Hematol. 2019 Aug;94(8):E209-E213. doi: 10.1002/ajh.25505. Epub 2019 May 21. No abstract available. PMID 31056762
- [Result] Baird JH, Frank MJ, Craig J, Patel S, Spiegel JY, Sahaf B, Oak JS, Younes SF, Ozawa MG, Yang E, Natkunam Y, Tamaresis J, Ehlinger Z, Reynolds WD, Arai S, Johnston L, Lowsky R, Meyer E, Negrin RS, Rezvani AR, Shiraz P, Sidana S, Weng WK, Davis KL, Ramakrishna S, Schultz L, Mullins C, Jacob A, Kirsch I, Feldman SA, Mackall CL, Miklos DB, Muffly L. CD22-directed CAR T-cell therapy induces complete remissions in CD19-directed CAR-refractory large B-cell lymphoma. Blood. 2021 Apr 29;137(17):2321-2325. doi: 10.1182/blood.2020009432. PMID 33512414
- [Result] Spiegel JY, Patel S, Muffly L, Hossain NM, Oak J, Baird JH, Frank MJ, Shiraz P, Sahaf B, Craig J, Iglesias M, Younes S, Natkunam Y, Ozawa MG, Yang E, Tamaresis J, Chinnasamy H, Ehlinger Z, Reynolds W, Lynn R, Rotiroti MC, Gkitsas N, Arai S, Johnston L, Lowsky R, Majzner RG, Meyer E, Negrin RS, Rezvani AR, Sidana S, Shizuru J, Weng WK, Mullins C, Jacob A, Kirsch I, Bazzano M, Zhou J, Mackay S, Bornheimer SJ, Schultz L, Ramakrishna S, Davis KL, Kong KA, Shah NN, Qin H, Fry T, Feldman S, Mackall CL, Miklos DB. CAR T cells with dual targeting of CD19 and CD22 in adult patients with recurrent or refractory B cell malignancies: a phase 1 trial. Nat Med. 2021 Aug;27(8):1419-1431. doi: 10.1038/s41591-021-01436-0. Epub 2021 Jul 26. PMID 34312556
- [Result] Cordoba S, Onuoha S, Thomas S, Pignataro DS, Hough R, Ghorashian S, Vora A, Bonney D, Veys P, Rao K, Lucchini G, Chiesa R, Chu J, Clark L, Fung MM, Smith K, Peticone C, Al-Hajj M, Baldan V, Ferrari M, Srivastava S, Jha R, Arce Vargas F, Duffy K, Day W, Virgo P, Wheeler L, Hancock J, Farzaneh F, Domning S, Zhang Y, Khokhar NZ, Peddareddigari VGR, Wynn R, Pule M, Amrolia PJ. CAR T cells with dual targeting of CD19 and CD22 in pediatric and young adult patients with relapsed or refractory B cell acute lymphoblastic leukemia: a phase 1 trial. Nat Med. 2021 Oct;27(10):1797-1805. doi: 10.1038/s41591-021-01497-1. Epub 2021 Oct 12. PMID 34642489
- [Result] Shalabi H, Kraft IL, Wang HW, Yuan CM, Yates B, Delbrook C, Zimbelman JD, Giller R, Stetler-Stevenson M, Jaffe ES, Lee DW, Shern JF, Fry TJ, Shah NN. Sequential loss of tumor surface antigens following chimeric antigen receptor T-cell therapies in diffuse large B-cell lymphoma. Haematologica. 2018 May;103(5):e215-e218. doi: 10.3324/haematol.2017.183459. Epub 2018 Feb 1. No abstract available. PMID 29419431
- [Result] Plaks V, Rossi JM, Chou J, Wang L, Poddar S, Han G, Wang Z, Kuang SQ, Chu F, Davis RE, Vega F, Bashir Z, Jacobson CA, Locke FL, Reagan PM, Rodig SJ, Lekakis LJ, Flinn IW, Miklos DB, Bot A, Neelapu SS. CD19 target evasion as a mechanism of relapse in large B-cell lymphoma treated with axicabtagene ciloleucel. Blood. 2021 Sep 23;138(12):1081-1085. doi: 10.1182/blood.2021010930. No abstract available. PMID 34041526